CLINICAL TRIAL: NCT00490607
Title: A Prospective Study Comparing the Incidence of Infantile Hemangiomas Following Normal Pregnancies Versus Pregnancies Complicated by Placental Abnormalities
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Rady Children's Hospital, San Diego (Other)
Other Study IDs: Hemangioma Study
Record Dates: First submitted 2007-06-21; First posted 2007-06-25 (Estimated); Last update posted 2007-06-25 (Estimated); Status verified 2007-06

CONDITIONS: Hemangioma
Keywords: Hemagiomas of infancy
MeSH Terms: conditions — Hemangioma

STUDY DESIGN:
Observational Model: Defined Population | Time Perspective: Prospective

SUMMARY:
The purpose of this study is to investigate the pathogenesis of hemangiomas of infancy as they relate to normal pregnancies and those pregnancies complicated by placenta abnormalities. Women of all gestational ages will be enrolled in the study. Maternal serum, placental, and cord blood samples will be obtained for each subject. A medical history will be obtained for each subject. Post-delivery a member of the study team will perform a cutaneous exam of the infant to establish what birthmarks are present at birth. Mother will receive four phone call follow ups to determine if the infant has had any skin changes. If yes, mother will be asked to bring the child in for evaluation. If a hemangioma is diagnosed, a blood draw will be performed.

ELIGIBILITY:
Inclusion Criteria:

* pregnant women delivering at Sharp Mary Birch Hospital for Women in San Diego, CA

Sex: Female
Age Groups: Child, Adult, Older Adult

CONTACTS AND LOCATIONS:
Overall Officials: Sheila F Friedlander, MA, Principal Investigator — Rady Children's Hospital, San Diego
Locations (1):
- Sharp Mary Birch Hospital for Women, San Diego, California, United States